CLINICAL TRIAL: NCT02737761
Title: Developing a Positive Psychology Intervention to Promote Health Behaviors in Heart Failure: Qualitative Research Phase
Brief Title: Researching Emotions And Cardiac Health
Acronym: REACH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Christopher Celano, Instructor in Psychiatry, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015P000069; 1K23HL123607-01A1 (NIH)
Record Dates: First submitted 2016-04-05; First posted 2016-04-14 (Estimated); Last update posted 2016-10-27 (Estimated); Status verified 2016-10

CONDITIONS: Congestive Heart Failure; Emotions; Patient Compliance
Keywords: Heart Failure; Positive Psychology; Adherence to Health Behaviors
MeSH Terms: conditions — Heart Failure; Patient Compliance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Optimal Adherence (Experimental): Participants will all undergo a qualitative interview and adherence measurements at baseline and 12 weeks after hospital discharge.
  In person the participants will receive a MEMSCaps device and an Actigraph accelerometer. They will be asked to begin wearing the accelerometer after their initial interview and to begin using the MEMSCaps device once they arrive at home. Participants will use the MEMSCap throughout the entire study and will wear the Actigraph for 2 weeks at baseline and again at 12 weeks.
  Interventions: Behavioral: Qualitative Interview and Adherence Measurements

INTERVENTIONS:
Behavioral: Qualitative Interview and Adherence Measurements — Subjects will undergo an open-ended, semi-structured interview within two weeks of enrollment. The interview will be approximately 1 hour in length, performed by study staff who have been trained in qualitative research methods. This interview will be completed again 12 weeks later. Subjects will complete the MOS SAS, Automated Self-Administered 24-hour recall (ASA24), Life Orientation Test-Revised (LOT-R), Positive and Negative Affect Schedule (PANAS), Hospital Anxiety and Depression Scale (HADS), Kansas City Cardiomyopathy Questionnaire (KCCQ), and Medical Outcomes Study Short Form-12 (SF-12) at baseline and again at 12 weeks.

SUMMARY:
The purpose of the study is to understand how positive emotions (e.g., optimism, happiness) are associated with health behavior adherence in patients with heart failure (HF), as well as whether performing exercises to improve positive emotions may help to improve health behavior adherence as well.

DETAILED DESCRIPTION:
The investigators are proposing a study that will specifically and innovatively focus on the development of a novel positive psychology intervention that is adapted for patients with HF. The MGH inpatient units and MGH Heart Center outpatients will serve as the source of subjects for the study, with patients who have a diagnosis of HF serving as potential subjects. The investigators will interview 30 HF patients within two weeks of enrollment in the study, and again three months later.

In this project, the investigators hope to do the following:

1. Identify, through qualitative research, deficits in positive emotional and cognitive states in clinically stable patients with New York Heart Association (NYHA) class II or III HF.
2. Examine potential links between positive emotional deficits and impaired health behaviors (low sodium diet, physical activity, medication adherence), as well as links between positive emotional sufficiency and successful health behaviors.
3. Identify other barriers to health behavior completion.
4. Explore strategies to enhance positive emotional and cognitive states in HF patients and inquire about the utility of potential PP exercises in these patients.
5. Develop a preliminary PP-based intervention using the above information.
6. Assess the feasibility of our proposed survey-based measures for adherence, psychological health, and physical health in this group of patients.
7. Explore the feasibility of using methods to objectively measure medication adherence and physical activity (via electronic pillcaps and accelerometers, respectively) in this population.

Baseline information about enrolled participants will be obtained from the patients, care providers, and the electronic medical record as required for characterization of our population. This information will include data regarding medical history (history of prior acute coronary syndrome, coronary artery bypass graft, congestive HF, hypertension, diabetes mellitus, hyperlipidemia, and current smoking), current medical variables (renal function, left ventricular ejection fraction, NYHA class), medications, and sociodemographic data (age, gender, race/ethnicity, living alone).

Participants will undergo an open-ended, semi-structured interview within 2 weeks of enrollment. The interview will be approximately 1 hour in length, performed by study staff who have been trained in qualitative research methods. Participants will then undergo another qualitative interview and repeat the battery of questionnaires again at 12 weeks.

Participants will wear an Actigraph accelerometer for 2 weeks at Baseline and again at 12 weeks to measure physical activity, and will also use a MEMSCap electronic pill counter throughout the study to measure medication adherence, respectively.

ELIGIBILITY:
Inclusion Criteria:

• Adult patients with NYHA class II or III HF admitted to an MGH inpatient unit or outpatients at the MGH Heart Center. Investigators will enroll subjects who develop mild to moderate HF symptoms during activity but not at rest. NYHA class II/III HF patients comprise the majority of subjects in studies that identify links between physical activity and improved exercise capacity, QoL, and survival making them an ideal study population. HF diagnosis, clinical stability, and NYHA class will be clarified with the inpatient or outpatient cardiology team.

Exclusion Criteria:

* Cognitive deficits impeding a subject's ability to provide informed consent or participate, assessed via a 6-item cognitive test that is sensitive and specific for screening for cognitive impairment in research subjects.
* Medical conditions precluding interviews or likely to lead to death within 6 months.
* Inability to speak English, inability to read or write, inability to walk, or lack of a telephone.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-01; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Themes related to how deficits in positive emotional states are associated with health behavior adherence | Qualitative data collected at Baseline
  Subjects will complete a structured interview at baseline, providing information about their own positive emotional states, identifying strategies to enhance positive emotions, linking the presence of positive emotions to better adherence to health-related behaviors, and identifying additional barriers (e.g., logistic, financial) to completing such behaviors.

SECONDARY OUTCOMES:
Changes in PANAS Scores | Baseline, 12 weeks
  The positive affect items on the Positive and Negative Affect Schedule (PANAS), a well-validated scale used in other intervention trials and in patients with HF, will be used to measure positive affect.
Changes in LOT-R Scores | Baseline, 12 weeks
  Life Orientation Test-Revised is a well-validated 6-item instrument used to measure dispositional optimism.
Changes in HADS Scores | Baseline, 12 weeks
  The Hospital Anxiety and Depression Scale will be used to measure depression and anxiety. This is a well-validated scale with few somatic symptom items that can confound mood/anxiety assessment in medically-ill patients.
Changes in KCCQ Scores | Baseline, 12 weeks
  The Kansas City Cardiomyopathy Questionnaire is a well-validated questionnaire of health status in HF. The full scale will be used to measure HF-specific health-related QoL (HRQoL), and an eight-question subset of the KCCQ will be used as a measure of HF symptoms.
Changes in SF-12 Scores | Baseline, 12 weeks
  The Medical Outcomes Study Short Form-12 (SF-12) will be used to measure quality of life. This is an instrument which has been used in multiple cardiac studies in the past.
Changes in MOS SAS Scores | Baseline, 12 weeks
  Three Medical Outcomes Study Specific Adherence Scale (MOS SAS) items assessing medication, diet, and exercise, will be measured individually and as a composite score.
Changes in daily sodium intake (as measured with the ASA24) | Baseline, 12 weeks
  The Automated Self-administered 24-hour recall (ASA24) is an online assessment tool based on the U.S. Department of Agriculture's (USDA) Automated Multi-Pass Method (AMPM). It will be used to calculate daily sodium intake.
Medication Adherence (MEMSCaps) | 12 weeks
  The MEMSCap has been used in patients with HF and is the most prevalent system for measuring adherence to PO medications. Investigators will measure adherence to a once-daily prescribed medication (aspirin, thiazide diuretic, statin, ACE inhibitor, or another once-daily cardiac medication, chosen in that order). Data will be continuously collected, and adherence noted by presence of bottle opening each day. Participants will use the pill counter throughout the study.
Physical Activity Adherence (Actigraph) | 12 weeks
  ActiGraph GT3X+ step counters are validated as measures of physical activity and have been used in numerous studies of physical activity in patients with medical illness. In this trial, participants will wear the accelerometer to assess the feasibility of doing so and to ensure adequate capture of physical activity.
Feasibility of MEMSCaps | Baseline and 12 weeks
  Feasibility will be measured by examining the rates of use of the MEMSCap.
Feasibility of Actigraph | Baseline and 12 weeks
  Feasibility will be measured by examining the rates of use of the Actigraph.
Themes related to how deficits in positive emotional states are associated with health behavior adherence at 12 weeks | Qualitative data collected at 12 weeks
  Subjects will complete a structured interview at 12 weeks, providing information about their own positive emotional states, identifying strategies to enhance positive emotions, linking the presence of positive emotions to better adherence to health-related behaviors, and identifying additional barriers (e.g., logistic, financial) to completing such behaviors.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher M Celano, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No